CLINICAL TRIAL: NCT02209701
Title: A Phase I Intensive Pharmacokinetic Study of Porfiromycin in Head and Neck Cancer and Other Cancer Patients With Solid Tumors Who Receive Radiation Therapy
Brief Title: Pharmacokinetic Study of Porfiromycin in Head and Neck Cancer and Other Cancer Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1164.3
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Porfiromycin

ARMS (1):
- Porfiromycin (Experimental)
  Interventions: Drug: Porfiromycin

INTERVENTIONS:
Drug: Porfiromycin

SUMMARY:
Study to determine the steady-state pharmacokinetics and urinary excretion of porfiromycin and major metabolites in head and neck cancer and other cancer patients with solid tumors who receive radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven advanced head and neck cancer or other solid tumors undergoing radiation therapy
* Patients with prior chemotherapy will be considered if chemotherapy occurred more than 30 days prior to this study
* Patients must be receiving concomitant radiotherapy (RT)
* Performance status of ≥ 70% on the Karnofsky performance scale (KPS)
* Must be ≥ 18 years of age
* Expected survival of at least three months
* Written informed consent

Exclusion Criteria:

* Patients who meet any of the following clinical laboratory criteria:

  * Granulocyte count of < 2000/mm**3
  * Platelets < 75,000/mm**3
  * Serum creatinine > 1.5 times the upper limit of normal
  * Bilirubin > 1.5 times the upper limit of normal
  * Prothrombin time and partial thromboplastin time > 1.5 times the upper limit of normal
* Women who are pregnant
* Men and women of child-bearing potential who are unwilling to utilize a medically acceptable method of contraception
* Patients who have any known bleeding disorder at the discretion of the investigator
* Presence of any other life-threatening illness, such as unstable angina, severe oxygen dependent chronic obstructive pulmonary disease, or unstable liver or renal disease
* Treatment with granulocyte colony-stimulating factor, granulocyte-macrophage colony-stimulating factor or Interleukin-1l within 30 days prior to the start of RT
* Patients who have had prior exposure to mitomycin C or porfiromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1999-12; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Assessment of serum concentrations of the analyte | up to 6 hours after drug infusion
Amount of analyte excreted in urine | 0-3 and 3-6 hours after infustion